CLINICAL TRIAL: NCT02794389
Title: How do Glutathione Levels Affect Compulsivity? A Double-blind, Placebo-controlled Study
Brief Title: Glutathione Levels and Compulsivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R44271/RE001
Record Dates: First submitted 2016-05-12; First posted 2016-06-09 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-02

CONDITIONS: Anorexia Nervosa; Compulsive Behavior
Keywords: Acetylcysteine
MeSH Terms: conditions — Anorexia Nervosa; Compulsive Behavior | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-acetyl cysteine (Experimental): 1200mg for 2 days 2400mg for 7 days
  Interventions: Drug: N-acetyl cysteine
- Placebo (Placebo Comparator): Magnesium stearate capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetyl cysteine
  Arms: N-acetyl cysteine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The investigators will examine whether compulsivity in those who score above-average (but below clinical cut-off) on an eating disorder questionnaire can be altered by 9 days of N-acetyl cysteine (NAC). N-acetyl cysteine has been shown to be of some benefit in individuals with other compulsive disorders, such as trichotillomania and addiction, so this research investigates whether a short period of time taking N-acetyl cysteine changes compulsivity, measured using cognitive tasks and questionnaires.

DETAILED DESCRIPTION:
Anorexia nervosa is a psychiatric disorder with a high mortality rate and for which there is very little evidence for pharmacological interventions of value. The picture is similar in bulimia nervosa, with a high mortality rate and with mixed outcomes from studies testing Selective Serotonin Reuptake Inhibitors (SSRIs). It is possible to conceptualise eating disorders as akin to compulsive disorders, especially noting that repetitive weighing, calorie counting and compulsive exercise and compensatory mechanisms might fit into a hypothetic obsessive-compulsive spectrum (OC spectrum). Some disorders on this OC spectrum are associated with oxidative stress. This may also be true in eating disorders: it has recently been found in a meta-analysis that there is evidence of increased oxidative stress markers in AN.

Glutathione is the main cellular anti-oxidant in mammals and it is possible to increase glutathione levels (and thus potentially combat oxidative stress) with a dietary supplement called N-Acetyl Cysteine (NAC). NAC is an acetylated form of the naturally occurring amino acid cysteine, and is converted to cysteine in the body. Cysteine is a key precursor of glutathione. Oral administration of cysteine itself does not increase brain glutathione levels because cysteine is poorly absorbed from the gastro-intestinal tract. However NAC is bioavailable and thus administration of it does increase glutathione in the brain.

Using NAC to increase glutathione levels has been shown to be beneficial in some compulsive disorders such as addictions, Obsessive-Compulsive Disorder (OCD) and related disorders such as trichotillomania in preliminary studies. There have been positive indications for use and evidence in pathological gambling, trichotillomania, OCD and cocaine addiction. However, NAC has not to our knowledge ever been considered for the treatment of eating disorders. This research therefore aims to investigate whether increasing glutathione can reduce neuropsychological markers of compulsivity in a group at risk for eating disorders.

The researchers have chosen to use a female non-patient group which is thought to be highly compulsive, but which will also be without the possible confounds of medication (as in OCD or addiction disorders) and without malnutrition (as in clinical eating disorders). Those recruited will be females, because there is evidence that there may be different risk factors and thus mechanisms underlying the development of eating disorders in males and females, such that recruiting both might produce a confound. The investigators have also chosen to use a short duration of NAC administration. This not only allows the use of a cross-over design without fears of high attrition rates and non-compliance, but it also will allow the detection of subtle and early changes in compulsivity. The hypothesis is thus that improvements will be seen in tasks measuring compulsivity, and also potentially in tasks which measure related constructs such as impulsivity, habit-based learning, and delay discounting. The researchers do not expect improvement in self-report symptom questionnaires. However, a possible future study would be a randomized clinical trial looking at increasing glutathione in a clinical group over time and how it affects clinical symptomatology.

The questionnaires chosen will identify eating disorder symptom levels (the Eating Attitudes Test - 26 (EAT-26) is a validated way of doing this) and look at compulsive starvation using the self-starvation scale (Godier & Park 2015). The Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders-IV (SCID) will be used to rule out those with a current Axis I diagnosis including an eating disorder, to prevent the complications of starvation and medication in this initial pilot study. The Eysenck Personality Questionnaire (EPQ) will be used to ascertain personality traits, and the National Adult Reading Test (NART) will be used to estimate Intelligence Quotient (IQ).

The rationale for choosing the tasks was based on the hypothesis that compulsivity may be improved by increasing glutathione levels. Thus, the tasks chosen are designed to pick up differences in different facets of compulsivity. The Wisconsin Card Sorting Task (WCST) is able to quantitatively measure set shifting, which is known to be impaired in eating disorders (Roberts et al. 2007) and is a facet of compulsivity. The Affective Go/No go picks up on attention bias within the umbrella of compulsivity; and the Attention Switching task picks up the ability to switch attention between different task demands, within the same compulsivity umbrella. The Cambridge Gambling Task is a good measure of disadvantageous decision making within the umbrella of impulsivity (which is thought to be orthogonally related to, rather than opposite to, compulsivity) (Fineberg et al. 2014). The sequential learning task has been used in OCD, where it is able to disentangle goal-directed learning from habitual learning based on two computational algorithms. The hypothesis is that compulsivity is related to a disturbance in goal-directed learning, with habit learning preferred leading to rigid behaviours (Gillan & Robbins 2014) (Voon et al. 2015). Thus it will be useful to see if more goal-directed and less habit learning occurs after increases in glutathione levels. The delay discount task measures the ability to ignore delays in time when considering reward value, which is relevant in eating disorders as often delay discounting is reduced so performance is better (Steinglass et al. 2012). This has an interesting interaction with impulsivity as it seems almost to be opposite to it, yet anorexic patients have shown a better performance. Thus this task might be useful as an exploratory measure. The Facial Expression Recognition Task (FERT) is very sensitive to early changes in emotional biases after only small pharmacological changes, and as the profile of individuals high eating disorder symptoms is different in this task compared to healthy controls (Jones et al. 2008) - it can operate as a positive control to identify if increased glutathione is having any effect on general emotional biases, even if it is not on compulsivity.

Because the aim of the study is to see whether NAC may lower compulsivity by increasing glutathione levels, a researcher will take a small venous blood sample (5mls) and a saliva sample prior to testing in both arms of the study to check to what to what extent NAC treatment elevates glutathione levels over placebo. Participants who do not wish to give blood will not be excluded but asked to provide a saliva sample only. Blood and saliva will be rendered acellular by centrifugation and stored until assay in the University Departments of Chemistry and Pharmacology. Once assayed any remaining sample will be discarded according to Standard Operating Procedures for sample disposal.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Females aged 18 to 40 years.
* Score between 9 and 19 on the EAT-26.
* Participant is a fluent English speaker

Exclusion Criteria:

* Any current psychotropic medications.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the study.
* BMI below 18.5, indicating that they are underweight.
* Any Axis I psychiatric disorder.
* History of allergies to drugs or vaccines or any component of the NAC or placebo capsule (gelatine, magnesium stearate, NAC).
* Pregnant, could be pregnant, breast feeding, or high risk of pregnancy (no reliable contraception use but sexual activity).
* Has taken part in a psychological or medical experiment involving taking any kinds of drugs within the last 6 weeks.
* Has had recent surgery.
* Taking selenium, vitamin E, or NAC.
* Current regular cigarette smoking of over 5 cigarettes per day.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in scores on the Berg Card-Sort Task (a measure of set-shifting) when taking N-acetyl cysteine compared to placebo | Change between study visit on the 9th day of taking NAC, and the study visit on the 9th day of taking placebo.
  Improvement in scores on the Berg Card-Sort Task (a version of the Wisconsin Card Sorting Task) after NAC compared to placebo. Analyse using paired-sample t-tests on the perseverative error totals for each participant at each visit.

SECONDARY OUTCOMES:
Change in scores on the Attention Switching Task when taking N-acetyl cysteine compared to placebo. | Change between study visit on the 9th day of taking NAC, and the study visit on the 9th day of taking placebo.
  Improvement in scores on the Attention Switching Task after NAC compared to placebo. Analyse using paired-sample t-tests.
Change in score on the Affective Go/No-Go task (measuring attentional bias) when taking N-acetyl cysteine compared to placebo | Change between study visit on the 9th day of taking NAC, and the study visit on the 9th day of taking placebo.
  Improvement in scores on the Affective Go/No-Go task after NAC compared to placebo. Analyse using paired-sample t-tests.
Change in scores on the Cambridge Gambling Task (measuring disadvantageous decision-making) when taking N-acetyl cysteine compared to placebo | Change between study visit on the 9th day of taking NAC, and the study visit on the 9th day of taking placebo.
  Change in scores on the Cambridge Gambling Task after NAC compared to placebo. Compare scores using paired-sample t-tests.
Change in sequential learning task score (a measure of excessive habit-learning) when taking N-acetyl cysteine compared to placebo. | Change between study visit on the 9th day of taking NAC, and the study visit on the 9th day of taking placebo.
  Improvement in scores on the sequential learning task after NAC compared to placebo. Analyse by comparing beta weight of interaction effect between groups (NAC and placebo).
Change in scores on delay discounting task when taking N-acetyl cysteine compared to placebo. | Change between study visit on the 9th day of taking NAC, and the study visit on the 9th day of taking placebo.
  Change in scores on the delay discounting task after NAC compared to placebo. Analyse using paired-sample t-tests.
To examine whether mood symptoms as indexed by the Hospital Anxiety and Depression Scale (HADS) change between baseline, N-acetyl cysteine administration and placebo administration. | Change between screening visit, study visit on the 9th day of taking N-acetyl cysteine, and the study visit on the 9th day of taking placebo.
  Examine scores on HADS and see if they change over those 3 timepoints. Use paired-sample t-tests on the total score on the questionnaire. May also separate the sub-scales for anxiety and depression and perform paired t-tests on these too, if thought necessary.
To examine whether eating disorder symptoms indexed by the EAT-26 change between baseline, N-acetyl cysteine administration, and placebo administration. | Change between screening visit, study visit on the 9th day of taking N-acetyl cysteine, and the study visit on the 9th day of taking placebo.
  Examine scores on EAT-26 and see whether they change over those 3 timepoints. Use paired-sample t-tests.
Examine change in score on the FERT when taking N-acetyl cysteine compared to placebo. | After 9 days of taking N-acetyl cysteine and after 9 days of taking placebo.
  Change in performance on the FERT, analysed using an ANOVA to investigate whether there is an interaction effect in accuracy between emotion recognition and group (N-acetyl cysteine, placebo).
Identify any difference in the side effect profile recorded daily during N-acetyl cysteine administration and placebo administration. | After 9 days of taking N-acetyl cysteine and after 9 days of taking placebo.
  Significantly greater scores on side effect questionnaire during 9 days of NAC vs. placebo. Scores will be derived by totalling all side effects from all 9 days of each arm, with absent corresponding to a score of 0, mild corresponding to a score of 1, moderate corresponding to a score of 2, severe corresponding to a score of 3.
Calculate the percentage of participants who correctly guess which treatment group they are in (N-acetyl cysteine vs. placebo). | After 9 days of taking NAC and placebo for each participant.
  Examine the guesses made as to whether NAC/placebo was taken, and calculate percentages correct.

CONTACTS AND LOCATIONS:
Overall Officials: Phil J Cowen, Prof, Principal Investigator — University of Oxford
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grant JE, Odlaug BL, Kim SW. A double-blind, placebo-controlled study of N-acetyl cysteine plus naltrexone for methamphetamine dependence. Eur Neuropsychopharmacol. 2010 Nov;20(11):823-8. doi: 10.1016/j.euroneuro.2010.06.018. Epub 2010 Jul 22. PMID 20655182
- [Background] Grant JE, Kim SW, Odlaug BL. N-acetyl cysteine, a glutamate-modulating agent, in the treatment of pathological gambling: a pilot study. Biol Psychiatry. 2007 Sep 15;62(6):652-7. doi: 10.1016/j.biopsych.2006.11.021. Epub 2007 Apr 18. PMID 17445781
- [Background] Grant JE, Fineberg N, van Ameringen M, Cath D, Visser H, Carmi L, Pallanti S, Hollander E, van Balkom AJ. New treatment models for compulsive disorders. Eur Neuropsychopharmacol. 2016 May;26(5):877-84. doi: 10.1016/j.euroneuro.2015.11.008. Epub 2015 Nov 18. PMID 26621260
- [Background] Gillan CM, Kosinski M, Whelan R, Phelps EA, Daw ND. Characterizing a psychiatric symptom dimension related to deficits in goal-directed control. Elife. 2016 Mar 1;5:e11305. doi: 10.7554/eLife.11305. PMID 26928075
- [Background] Gillan CM, Otto AR, Phelps EA, Daw ND. Model-based learning protects against forming habits. Cogn Affect Behav Neurosci. 2015 Sep;15(3):523-36. doi: 10.3758/s13415-015-0347-6. PMID 25801925
- [Background] Voon V, Derbyshire K, Ruck C, Irvine MA, Worbe Y, Enander J, Schreiber LR, Gillan C, Fineberg NA, Sahakian BJ, Robbins TW, Harrison NA, Wood J, Daw ND, Dayan P, Grant JE, Bullmore ET. Disorders of compulsivity: a common bias towards learning habits. Mol Psychiatry. 2015 Mar;20(3):345-52. doi: 10.1038/mp.2014.44. Epub 2014 May 20. PMID 24840709
- [Background] Godier LR, Park RJ. Compulsivity in anorexia nervosa: a transdiagnostic concept. Front Psychol. 2014 Jul 17;5:778. doi: 10.3389/fpsyg.2014.00778. eCollection 2014. PMID 25101036
- [Derived] Hoffman J, Williams T, Rothbart R, Ipser JC, Fineberg N, Chamberlain SR, Stein DJ. Pharmacotherapy for trichotillomania. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD007662. doi: 10.1002/14651858.CD007662.pub3. PMID 34582562